CLINICAL TRIAL: NCT04137562
Title: A Multicenter, Randomized, Single-Blind, Phase Ⅱ Clinical Trial and Open Label Long-term Observation Study of ADSTEM Inj. to Evaluate the Safety and Efficacy in Patients With Moderate to Severe Subacute and Chronic Atopic Dermatitis
Brief Title: Safety and Efficacy in Patients With Moderate to Severe Subacute and Chronic Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EHL Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-CP-18-1; 30902 (Other Grant/Funding Number: Republic of Korea Ministry of Food and Durg Safety)
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
Keywords: Adipose Derived Mesenchymal Stem cell; ADMSC; AD; Inflammatory disease; ADMC; Stem cell; ehlbio
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and efficacy outcome assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADSTEM Inj. (Experimental): ADSTEM Inj. hAD-MSC 1.0x10^8 cells
  Interventions: Biological: ADSTEM Inj.
- Placebo (Placebo Comparator): 0.9% Normal Saline Inj.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ADSTEM Inj. — Two 5mL of the following study drug is pre-mixed with 320mL of 0.9% normal saline is injected intravenously twice for the duration of the study. Treatment group: ADSTEM Inj. 0.5x10^8 cells/5mL
  Arms: ADSTEM Inj.
Other: Placebo — 330mL of 0.9% normal saline is injected intravenously twice for the duration of the study.
  Arms: Placebo

SUMMARY:
A Multicenter, Randomized, Single-Blind, Phase Ⅱ Clinical Trial and Open Label Long-term Observation Study of ADSTEM Inj. to Evaluate the Safety and Efficacy in Patients with Moderate to Severe Subacute and Chronic Atopic Dermatitis.

The aim of this study is to evaluate the safety and efficacy of ADSTEM Inj. against Placebo in the treatment of atopic dermatitis in patients with moderate to severe acute and chronic atopic.

DETAILED DESCRIPTION:
This clinical trial is designed with multi-organization, random assignment, single-blind, second-phase clinical trials and open long-term follow up studies, and is intended for patients with secondary or above subacuteal and chronic atopic dermatitis. If the test subjects voluntarily agree in writing to participate in this clinical trial, they shall conduct the examination and examination required for four weeks prior to administration of the investigational product (visit 1) in accordance with the clinical trial plan. As a result of the suitability assessment of the test subjects, those who comply with the inclusion/exclusion criteria, adipose tissue will be collected through the liposuction method and randomly assigned to each arms. Subjects who are eligible for administration of the investigational product on the day of administration (visit 2) under the investigator's judgment are given intravenous administration of the clinical trial medication once at the date of administration (visit 2, visit 3) and follow-up inspection is conducted at 4 weeks, 8 weeks, 12 weeks, and 16 weeks after the first administration of the investigational product and safety and efficacy assessments are conducted for a total of 16 weeks. The test subjects assigned to the placebo group shall be compensated by administering a experimental drug on demand after the visit 6. It is a principle to administer the test drug prepared from the previously obtained adipose tissue, and it is possible to carry out further adipose tissue collection if necessary. However, no safety and efficacy assessments of compensatory treatments will be collected. Safety and efficacy will be analyzed after all the subjects has completed visit 6. For the experimental group only, long-term observation study for safety assessment is conducted at the point of 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 48 months, and 60 months after the second administration of the investigational product for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* At the time of visit 1, only men and women aged between 19 and 70
* Patients with atopic dermatitis meeting the Hanifin and Rajka diagnostic criteria
* Subacute and chronic patients with symptoms of atopic dermatitis lasting at least 6 months
* Patients with moderate to severe atopic dermatitis who meet all of the following criteria

  1. SCORAD score ≥ 20points
  2. EASI score ≥ 12points
  3. BSA ≥ 10%
* Patients with inadequate response to the stable use of topical atopic dermatitis treatment within 24 weeks prior to study initiation, or those who are unable to administer topical atopic dermatitis treatment due to safety reasons
* Patients who voluntarily agreed in writing to participate in this clinical trial

Exclusion Criteria:

* Patients with systemic infection symptoms at the time of clinical trials
* Patients with HIV, HBV, HCV, Syphilis test positive
* Patients with uncontrolled asthma disease at the time of clinical trial participation
* Patients who were considered inevitable to receive the medication from 1 month prior to administration of the clinical trial drug to visit 6 such as Immune function modifier(tacrolimus, pimecrolimus, cyclosporine, etc.), and high-frequency topical steroids in Groups 1 to 5, systemic steroids, systemic photochemotherapy, medication that are thought to affect other immune functions (such as immunoglobulin therapy like dupilumab, tralloquinap and desensitization therapy, etc.)
* Women who are pregnant, breastfeeding or have a pregnancy plan up to visit 6 or who do not use available contraceptive methods (women of childbearing age must be negative in screening pregnancy test)
* If patients are the male subject, Those who do not agree to have a contraception during the clinical trial (If the male subject or female partner is infertile, the above-mentioned contravention method is unnecessary)
* Patients participating in other clinical trials or participating in other clinical trials within the last 30 days
* Patients who have experienced significant adverse events during treatment with stem cell therapies
* Patients with stem cell therapy doses or history of participating in clinical trials
* Patients with a history of hypersensitivity to antibiotics and antifungal agents used in the manufacture of medicines for clinical trials
* Patients with renal dysfunction whose creatinine level is more than twice the normal upper limit in the screening test
* Patients with hepatic dysfunction whose AST (Aspartate Amino Transaminase) and ALT (Alanine Amino Transaminase) levels are more than three times the normal upper limit
* Patients who are not suitable for this clinical trial under the judgment of the other examiners

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
EASI-50 | 16 weeks
  Percentage of subjects whose EASI score decreased by 50% or more at 16 weeks compared to baseline

SECONDARY OUTCOMES:
EASI-50 | 4, 8, 12 weeks
  Percentage of subjects whose EASI score decreased by 50% or more at 4, 8 and 12 weeks compared to baseline
EASI-75 | 4, 8, 12, 16 weeks
  Percentage of subjects whose EASI score decreased by 75% or more at 4, 8, 12 and 16 weeks compared to baseline
EASI score | 4, 8, 12, 16 weeks
  EASI score change at 4, 8, 12 and 16 weeks compared to baseline
SCORAD-50 | 4, 8, 12, 16 weeks
  Percentage of subjects whose SCORAD score decreased by 50% or more at 4, 8, 12 and 16 weeks compared to baseline
SCORAD-75 | 4, 8, 12, 16 weeks
  Percentage of subjects whose SCORAD score decreased 75% or more at 4, 8, 12 and 16 weeks compared to baseline
SCORAD score | 4, 8, 12, 16 weeks
  SCORAD score change at 4, 8, 12 and 16 weeks compared to baseline
SCORAD subgroup | 4, 8, 12, 16 weeks
  SCORAD evaluation items(Extent Criteria, erythema, edema/population, oozing/crusting, excoriation, lichenification, dryness, pruritus, insomnia) score change at 4, 8, 12 and 16 weeks compared to baseline
Severity | 4, 8, 12, 16 weeks
  Severity change of disease at 4, 8, 12 and 16 weeks compared to baseline
IGA grade | 4, 8, 12, 16 weeks
  Investigator's Global Assessment (IGA) score at 4, 8, 12 and 16 weeks compared to baseline
IGA -1 or more grade | 4, 8, 12, 16 weeks
  Percentage of subjects who dropped one or more grades on the Investigator's Global Assessment (IGA) score at 4, 8, 12 and 16 weeks compared to baseline
IGA -2 or more grade | 4, 8, 12, 16 weeks
  Percentage of subjects who dropped two or more grades on the Investigator's Global Assessment (IGA) score at 4, 8, 12 and 16 weeks compared to baseline
Total IgE | 4, 8, 12, 16 weeks
  Total IgE change at 4, 8, 12, 16 weeks compared to baseline
PGE2 and ECP | 4, 8, 12, 16 weeks
  Prostaglandin E2 (PGE2) and Eosinophil Cationic Protein (ECP) changes at 4, 8, 12 and 16 weeks compared to baseline
Immune cytokine | 4, 8, 12, 16 weeks
  TGF-1, interleukin (IL)-4, 5, 6, 8, 13, 31 and CCL17 at 4, 8, 12 and 16 weeks compared to baseline
Remedy used days and frequency | 4, 8, 12, 16 weeks
  Days and frequency of used remedies at 4, 8, 12 and 16 weeks
Remedy used subjects | 4, 8, 12, 16 weeks
  Percentage of subjects whom used remedies at 4, 8,12 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seongjun Seo, M.D, Ph.D, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Sanguk Son, M.D, Ph.D, Principal Investigator — Korea University Ansan Hospital; Soyeon Jo, M.D, Ph.D, Principal Investigator — SMG-SNU Boramae Medical Center; Young-joon Seo, M.D, Ph.D, Principal Investigator — Chungnam National University Hospital; Donghun Lee, M.D, Ph.D, Principal Investigator — Seoul National University Hospital; Mingyeong Shin, M.D, Ph.D, Principal Investigator — Kyunghee University Medical Center
Locations (6):
- South Korea (6):
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Korea University AnSan Hospital, Ansan, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul, Seoulteukbyeolsi
  - Kyunghee University Medical Center, Seoul, Seoulteukbyeolsi
  - Seoul National University Hospital, Seoul, Seoulteukbyeolsi
  - SMG-SNU Boramae Medical Center, Seoul, Seoulteukbyeolsi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seok J, Kim SY, Lee WG, Shin MK, Lee DH, Seo YJ, Cho S, Park KY, Son SW, Lee SH, Seo JS, Seo SJ. Efficacy and safety of autologous adipose-derived stem cells in subjects with moderate to severe atopic dermatitis: a multicenter, randomized, single-blind, placebo-controlled, phase 2 trial. Stem Cell Res Ther. 2025 Dec 2;16(1):671. doi: 10.1186/s13287-025-04763-y. PMID 41331725